CLINICAL TRIAL: NCT05771155
Title: A Randomized, Double-blind, Multicenter Phase 3 Study in Patients With Moderately to Severely Active Ulcerative Colitis (UC) to Compare the Efficacy, Safety and Immunogenicity of PB016 and Entyvio® for the Induction and Maintenance of Clinical Response and Remission
Brief Title: Efficacy, Safety and Immunogenicity of the Proposed Biosimilar Vedolizumab PB016 in Comparison With Entyvio®
Acronym: UCESIVE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Polpharma Biologics S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PB016-03-01
Record Dates: First submitted 2023-03-01; First posted 2023-03-16 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2024-07

CONDITIONS: Ulcerative Colitis
Keywords: ulcerative colitis; vedolizumab; biosimilar
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- PB016 (300 mg IV) (Experimental): PB016 will be administered to patients with moderately to severely active UC on Weeks 0, 2 and 6, and once every 8 weeks thereafter, per the approved dosing regimen of Entyvio®
  Interventions: Biological: Intravenous (IV) infusions
- Entyvio® (300 mg IV) (Active Comparator): Entyvio® will be administered to patients with moderately to severely active UC on Weeks 0, 2 and 6, and once every 8 weeks thereafter, per the approved dosing regimen of Entyvio®
  Interventions: Biological: Intravenous (IV) infusions

INTERVENTIONS:
Biological: Intravenous (IV) infusions — Intravenous (IV) infusions of a dose of 300mg, on Weeks 0, 2 and 6, 14, 22, 30, 38 and 46

SUMMARY:
This is a multi-center, randomized, parallel arm, double-blind study with approximately 750 participants with moderately to severely active Colitis Ulcerosa randomized to receive either PB016 or Entyvio®

DETAILED DESCRIPTION:
This is a multi-center, randomized, parallel arm, double-blind study with a total duration of 54 weeks. Approximately 750 participants with moderately to severely active Colitis Ulcerosa will be randomized to receive up to eight doses of either PB016 or Entyvio®.

The study will be conducted at up to 200 study centers, located in approximately 18 countries worldwide.

The clinical trial is designed to compare the efficacy, safety, and immunogenicity of 300 mg IV PB016 versus Entyvio® in patients with moderately to severely active UC.

The active period of Study PB016-03-01 comprises the following:

* Stage 1: Induction Period - after 1:1 randomization, intravenous infusions of either PB016 or Entyvio® at a dose of 300 mg at Weeks 0 and 2.
* Stage 2: Maintenance Period - further doses at Weeks 6, 14, 22, 30, 38, and 46.
* Stage 3: Follow-up Period - At Week 54, a safety follow-up call will be conducted.

ELIGIBILITY:
(Selected) Inclusion Criteria:

* Age ≥18 and ≤75 years at Screening.
* At Screening, females of childbearing potential must be non-pregnant and non-lactating; or females should be of non-childbearing potential (either surgically sterilized or physiologically incapable of becoming pregnant, or at least 1 year post-menopausal [amenorrhea duration of 12 consecutive months]); non-pregnancy will be confirmed for all females of childbearing potential by a serum pregnancy test conducted at Screening.
* Female patients of childbearing potential, with a fertile male sexual partner, must use adequate contraception from Screening until 18 weeks after the last dose of study drug. Adequate contraception is defined as using hormonal contraceptives or an intrauterine device, combined with at least one of the following forms of contraception: a diaphragm or cervical cap, or a condom. Total abstinence from heterosexual activity, in accordance with the lifestyle of the patient, is acceptable.
* Male patients who are sexually active with women of childbearing potential agree they will use adequate contraception from Screening until 90 days after the last dose of study drug if not surgically sterilized at least 6 months before Screening (with a post-vasectomy semen analysis negative for sperm). Male patients must not donate sperm until 90 days after the last dose of study drug. Adequate contraception for the male patient and his female partner of childbearing potential is defined as using hormonal contraceptives or an intrauterine device, combined with at least one of the following forms of contraception: a diaphragm or cervical cap, or a condom. Total abstinence from heterosexual activity, in accordance with the lifestyle of the patient, is acceptable.
* Diagnosis of moderate to severe UC
* Evidence of UC extending proximal to the rectum (≥15 cm of involved colon).
* Patients with a family history of colorectal cancer, personal history of increased colorectal cancer risk, age >45 years, or other known risk factor must be up-to-date on colorectal cancer surveillance (may be performed during Screening).
* Demonstrated an inadequate response to, loss of response to, or intolerance to at least 1 of the following agents:

Corticosteroids, Immunomodulators, TNFα antagonists

* Able to participate in all aspects of this clinical study, including collection of tissue biopsies.
* Male or female patient who is voluntarily able to give informed consent.

(Selected) Exclusion Criteria:

* Previous exposure to vedolizumab (Entyvio® or any other investigational vedolizumab containing product).
* Female patients who are lactating or have a positive serum pregnancy test during the Screening Period or a positive urine pregnancy test on Day 0 prior to study drug administration.
* Has received any investigational or approved biologic or biosimilar agent within 60 days or 5 half-lives prior to randomization (whichever is longer).
* Evidence of abdominal abscess or toxic megacolon at the Screening Visit.
* Extensive colonic resection, subtotal or total colectomy.
* History of ileostomy, colostomy, or known fixed symptomatic stenosis of the intestine.
* History or evidence of colonic mucosal dysplasia.
* Diagnosis of Crohn's disease, microscopic colitis, ischemic colitis or indeterminate colitis.
* Had any surgical procedure requiring general anesthesia within 30 days prior to randomization or the patient currently requires or is anticipated to require surgical intervention for UC during the study.
* Has history or evidence of adenomatous colonic polyps that have not been removed, or colonic mucosal dysplasia.
* Has any of the following:

Evidence of a serious active or clinically significant infection requiring medical treatment or that in the opinion of the Investigator would confound the study results, during Screening or has been hospitalized or treated for such infection within 60 days of Baseline (e.g., sepsis, cytomegalovirus, listeriosis or opportunistic infections such as PML).

OR Evidence of or received treatment for C. difficile infection within 60 days, or other intestinal pathogen within 30 days prior to Screening. Rescreening of treated patients with no clinical signs and subsequent negative test results can be allowed at the Investigator's discretion.

OR Other current or recent (within 30 days prior to Screening) clinically significant infection (e.g., pneumonia, pyelonephritis).

* Chronic hepatitis B or C infection. Patients with positive viral serology at Screening for infection with hepatitis B (HBV), or hepatitis C virus (HCV) may be eligible if polymerase chain reaction test is negative, and the patient receives standard of care antiviral prophylaxis (if applicable).
* Known active TB.
* Has any identified congenital or acquired immunodeficiency (e.g., common variable immunodeficiency, human immunodeficiency virus [HIV] infection, organ transplantation).
* Has a history of hypersensitivity or allergies to the ingredients of Entyvio®.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2023-07-24 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
To demonstrate similarity of effect of induction treatment with IV formulations of PB016 and Entyvio® on clinical response rate at 6 weeks | Change from baseline to Week 6
  Clinical response rate, defined as the proportion of patients with a reduction in complete Mayo score

SECONDARY OUTCOMES:
To demonstrate similarity of effect of maintenance treatment with IV formulations of PB016 and Entyvio® on clinical response rate | Change from baseline to Week 52
  Clinical response rate at Week 52
To demonstrate similarity of effect of IV PB016 and Entyvio® on partial Mayo score | Change from baseline up to week 52
  Change from Baseline in partial Mayo score
To demonstrate similarity of effect of IV PB016 and Entyvio® on clinical remission rate | Change from baseline up to week 52
  Clinical remission rate
To demonstrate similarity of effect of IV PB016 and Entyvio® on mucosal healing rate | Change from baseline up to week 52
  Mucosal healing rate
To demonstrate similarity of effect of IV PB016 and Entyvio® on corticosteroid-free remission rate | Change from baseline to Week 52
  Corticosteroid-free remission rate, defined as the proportion of patients using oral corticosteroids at Baseline who have discontinued corticosteroids and are in clinical remission at Week 52
To compare the safety profiles of PB016 and Entyvio® | Change from baseline up to week 54
  * Number of patients with adverse events (AEs) and serious adverse events (SAEs)
  * Number of patients discontinuing treatment due to AEs or SAEs
To demonstrate similarity of IV PB016 and Entyvio® on immunogenicity | Change from baseline up to week 52
  Number of patients with anti-drug antibodies (ADAs) and neutralizing antibodies (NAb)

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Rethy, MD, Study Director — Polpharma Biologics S.A.
Locations (1):
- Todua Clinic LLC, Tbilisi, Georgia

IPD SHARING:
Plan to Share IPD: No